CLINICAL TRIAL: NCT00055510
Title: A Blinded Study Conducted at Multiple Centers Evaluating Various Doses of an Investigational Agent (BO-653) Against Placebo, for Safety and Effectiveness in Preventing Post-Angioplasty Blood Vessel Re-Closure (Restenosis) in Stented Vessels.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chugai Pharma USA (Industry)
Purpose: Treatment
Other Study IDs: BO-004
Record Dates: First submitted 2003-03-04; First posted 2003-03-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-02

CONDITIONS: Graft Occlusion, Vascular; Coronary Restenosis; Atherosclerosis
Keywords: BO-653; Coronary restenosis; Stent restenosis; LDL oxidative inhibitor; Antioxidant
MeSH Terms: conditions — Graft Occlusion, Vascular; Coronary Restenosis; Atherosclerosis | interventions — 2,3-dihydro-5-hydroxy-2,2-dipentyl-4,6-di-tert-butylbenzofuran

INTERVENTIONS:
Drug: BO-653

SUMMARY:
This research study is intended to evaluate the safety and effectiveness of 3 different doses of BO-653, an investigational inhibitor of LDL cholesterol oxidation, when given orally twice a day compared to placebo (an inactive substance) in preventing restenosis (closure of vessel) within six months after stent implantation. Patients must be enrolled into this study within 24 hours after the stenting procedure.

Additionally, over a 1- to 9-month post-stent period, the study will compare the safety and effectiveness of BO-653 versus placebo for measures of coronary artery vessel size by quantitative coronary angiography, major adverse cardiac events, and effects on the oxidative status of plasma lipids and other plasma components.

ELIGIBILITY:
Major Inclusion Criteria - Others Stipulated within the Protocol

The study physician must assure you:

* Are at least 18 years of age and have achieved a successful stent placement procedure as defined by ≤ 10% residual stenosis, no residual dissection, TIMI flow > 3 (complete perfusion), and lack of procedural coronary perforation utilizing an FDA-approved stent, excluding self-expanding, coil, polymer and pharmacologic coated (heparin OK) stents.
* Have at least one untreated target lesion in a native coronary artery meeting study entry criteria for diameter (≥ 2.5mm and ≤ 3.5mm), stenosis (≥ 50% and < 100%), and stent length (≥ 13mm and ≤ 36mm, or total of two stents ≤ 45mm).
* Have a documented history of angina pectoris or a positive functional study.
* Have no symptoms suggestive of an MI (heart attack) OR have cardiac isoenzymes (CK-MB) within normal range at least 24 hours prior to stent procedure.
* Use effective birth control measures, or are unable to conceive children.
* Are willing to have a repeat angiogram after 6 months.

Major Exclusion Criteria - Others Stipulated within the Protocol

The study physician must assure you:

* Have not had any coronary intervention within 30 days before, and for an expected 30 days after stenting.
* Have not had a cerebrovascular accident or transient ischemic attack within 90 days prior to stent placement.
* Have not had stent procedure as a bridge to non-emergency planned bypass.
* Have not had a stent placed within the target vessel less than 9 months ago, or less than 5mm from the closest edge of an adjacent lesion.
* Do not have an unprotected left main coronary artery disease.
* Do not have a left ventricular ejection fraction of < 30%.
* Do not have a target lesion that is located at the ostium (< 2mm from origin of left anterior descending, right coronary artery, or circumflex vessel), involves a side branch ≥2.0mm diameter, is moderately to severely calcified, or requires use of an atherectomy device.
* Have not had a heart transplant.
* Do not have a 12-lead ECG with a QTc interval pre- or post stent placement ≥ 460 msec (males), or ≥ 470 msec (females).
* Do not have any medical, surgical or psychiatric condition, or be medical unstable as would prevent you from safely participating in the trial.
* Do not have clinically relevant bleeding, clotting, or immune disorders or be intolerant of platelet inhibitors and/or anticoagulants.
* Are not taking rifampin, carbamazepine, phenobarbitol, cyclophosphamide, ifosfamide, artemisinin, mephenytoin, phenytoin, or cholestyramine.
* Have no clinically significant laboratory abnormality (specified: creatinine ≥ 2.2 mg/dl, liver function tests ≥ 2.0 times the upper limit of normal).
* Have not participated in any investigational study within past 30 days.
* Are not allergic or intolerant to soybean products.
* Are not taking vitamin E in excess of 150 I.U. per day and that you are unwilling to stop.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - St. Luke's Medical Center, Phoenix, Arizona
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Cardiovascular Associates of the Peninsula, Burlingame, California
  - Foundation for Cardiovascular Medicine, La Jolla, California
  - La Mesa Cardiac Center, La Mesa, California
  - Clinical Research Center of California, San Diego, California
  - Veterans Affairs Medical Center, San Diego, California
  - University of Florida Health Science Center, Jacksonville, Florida
  - Miami International Cardiology Consultants, Miami Beach, Florida
  - Mediquest Research Group, Ocala, Florida
  - Midwest Heart Research Foundation, Lombard, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Alton Ochsner Medical Foundation, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Borgess Medical Center, Kalamazoo, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - St. Louis University, St Louis, Missouri
  - Nevada Cardiology Associates, Las Vegas, Nevada
  - University of Rochester Medical Center, Rochester, New York
  - Asheville Cardiology Associates, PA, Asheville, North Carolina
  - Northwestern Memorial Hospital, Elyria, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Austin Heart, Austin, Texas
  - IRCI Institute for Research in Cardiovascular Interventions at The Methodist DeBakey Heart Center, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah